CLINICAL TRIAL: NCT01115920
Title: A Phase I Study in Healthy Male and Healthy Female Subjects to Characterize the Safety, Tolerability, and Pharmacokinetics of Intravenous Infusion of MTP-131 (Bendavia™) Using a Randomized, Double-Blind, Placebo-Controlled, Parallel Group Design
Brief Title: Study to Evaluate Safety, Tolerability, and Pharmacokinetics (PK) of Intravenous (IV) Infusion of MTP-131 (Bendavia™) in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stealth BioTherapeutics Inc. (Industry)
Responsible Party: Richard Straube, MD, Chief Medical Officer, Stealth Peptides, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPIRI-101
Record Dates: First submitted 2010-04-30; First posted 2010-05-04 (Estimated); Last update posted 2010-11-18 (Estimated); Status verified 2010-11

CONDITIONS: Healthy
Keywords: Drug Safety; Clinical Trial, Phase I; Nontherapeutic Human Experimentation; Heading Pharmacokinetics; Phase I Safety and Tolerability
MeSH Terms: interventions — arginyl-2,'6'-dimethyltyrosyl-lysyl-phenylalaninamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Arm 1 (Experimental): Cohort 1, Dose 0.010 mg/kg/hr Active (6), Placebo (2), Total Subjects (8)
  Interventions: Drug: MTP-131 (Bendavia™)
- Arm 2 (Experimental): Cohort 2, Dose 0.025 mg/kg/hr Active (6), Placebo (2), Total Subjects (8)
  Interventions: Drug: MTP-131 (Bendavia™)
- Arm 3 (Experimental): Cohort 3, Dose 0.050 mg/kg/hr Active (6), Placebo (2), Total Subjects (8)
  Interventions: Drug: MTP-131 (Bendavia™)
- Arm 4 (Experimental): Cohort 4, Dose 0.100 mg/kg/hr Active (6), Placebo (2), Total Subjects (8)
  Interventions: Drug: MTP-131 (Bendavia™)
- Arm 5 (Experimental): Cohort 5, Dose 0.250 mg/kg/hr Active (6), Placebo (2), Total Subjects (8)
  Interventions: Drug: MTP-131 (Bendavia™)

INTERVENTIONS:
Drug: MTP-131 (Bendavia™) — Single 4 hour intravenous infusion

SUMMARY:
This is the first study of MTP-131 (Bendavia™) in humans. The objective of this study is to evaluate the safety, tolerability, and pharmacokinetics of escalating single intravenous infusion doses of MTP-131.

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate the safety and tolerability of MTP-131 in healthy volunteers following a single intravenous infusion. The secondary objective is to evaluate the pharmacokinetics of MTP-131. This is a double-blind, placebo-controlled, randomized trial. A total of 40 eligible subjects will be enrolled and randomized in a 3:1 active to placebo ratio for a total of 5 treatment groups of 8 volunteers. As far as is logistically possible, each treatment group will have similar numbers of male and female volunteers. After the last subject for each cohort has completed the day 3 clinical assessment and no stopping rules have been met according to Safety Review Board decision, the next cohort will commence.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males or females age ≥18 years of age with signed informed consent.
* Women who are not post-menopausal or surgically sterile must have a negative serum pregnancy test at screening and within 24 hours of treatment and who agree to use effective contraception for 30 days following the study.

Exclusion Criteria:

* Clinically significant laboratory abnormalities,
* Clinically significant abnormalities on physical examination,
* BMI of less than 18 kg/m2 or greater than 32 kg/m2,
* Any disease or condition that might compromise the cardiovascular, hematological, renal, hepatic, pulmonary (including chronic asthma), endocrine (e.g., diabetes), central nervous, or gastrointestinal (including an ulcer) systems,
* History of seizures or epilepsy,
* History of serious mental illness,
* Participant in unrelated research involving investigational product within 30 days before planned date of drug administration,
* Positive serology for HIV 1, HIV 2, HBsAg, or HCV,
* Fever greater than 37.5°C at the time of planned dosing,
* Suspicion of or recent history of alcohol or substance abuse,
* Donated blood or blood products within the past 30 days,
* Women who are pregnant or breastfeeding,
* Employee or family member of the investigational site, and
* Subjects who currently smoke cigarettes, cigars, pipes or chew tobacco products,
* Subjects who are either unwilling to agree to refrain from use or found to be using:

  1. Alcohol, caffeine, xanthine-containing food or beverages, nicotine products and over-the-counter medications with the exception of Tylenol from 24 hours prior to dosing and throughout the confinement period
  2. Prescription medications from 14 days prior to and 7 days post treatment
  3. Oral contraceptives without concomitant use of double-barrier contraceptives (condom, diaphragm with spermicide) for a period of 7 days prior to and 30 days post treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-05; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Treatment emergent adverse events in treatment group versus placebo group | 7 days
  Safety assessments including vital signs, physical exam,12-lead ECG, serum chemistry, hematology, and urinalysis will be collected the day prior to and for 7 days following study drug infusion. These parameters will be assessed for clinically significant abnormalities.

SECONDARY OUTCOMES:
Pharmacokinetics of MTP-131 including Css, Cmax, tmax, t½, AUC and dose proportionality. | Pre-infusion through 32 hours post infusion
  Css (plasma steady state concentration), Cmax (observed peak plasma concentration), tmax (time of observed peak), AUC0-t (area under the plasma concentration time curve from time zero to the last quantifiable timepoint), AUC0-∞ (area under the plasma concentration time curve from time zero to infinity), λz (terminal [or elimination rate] phase rate constant), t½ (terminal half-life), CL (plasma clearance) and Vss (volume of distribution at steady state) will be determined for MTP-131. Ae (amount excreted in the urine) and CLr (renal clearance) may also be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Lasseter, MD, Principal Investigator — Clinical Pharmacology of Miami, Inc.
Locations (1):
- Clinical Pharmacology of Miami, Inc., Miami, Florida, United States